CLINICAL TRIAL: NCT00285207
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Trial of the Use of 4,4'-Dihydroxybenzophenone-2,4-Dinitrophenyl-hydrazone (A-007) Topical Gel in the Treatment of High-Grade Squamous Intraepithelial Lesions (HSIL) of the Cervix
Brief Title: Safety and Efficacy of A-007 Topical Gel in the Treatment of High-Grade Squamous Intraepithelial Lesions (HSIL) of the Cervix
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tigris Pharmaceuticals (Industry)
Responsible Party: Chief Medical Officer, Tigris
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG-001
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Results first posted 2010-10-11 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2010-09

CONDITIONS: Cervical Intraepithelial Neoplasia; Uterine Cervical Dysplasia
Keywords: Cervical Intraepithelial Neoplasia (CIN); High-grade Cervical Intraepithelial Neoplasia; High-grade Squamous Intraepithelial Lesions (HSIL); Human Papilloma Virus (HPV); High-Grade Cervical Intraepithelial Lesions (CIN 2/3)
MeSH Terms: conditions — Uterine Cervical Dysplasia; Squamous Intraepithelial Lesions | interventions — 4,4'-dihydroxybenzophenone-2,4-dinitrophenylhydrazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo administered topically to the cervix via intravaginal applicator for 5 consecutive days of a 28-day cycle for 2 cycles.
  Interventions: Drug: placebo
- A007 (Experimental): 0.25% A007 administered topically to the cervix via intravaginal applicator for 5 consecutive days of a 28-day cycle for 2 cycles.
  Interventions: Drug: A007

INTERVENTIONS:
Drug: placebo — 5 days of 28 day cycle for 2 cycles
  Arms: Placebo
Drug: A007 — 5 days of 28 day cycle
  Arms: A007

SUMMARY:
A-007 is an investigational therapy which may be effective in the treatment of pre-cancerous cervical dysplasia (abnormal cell growth). The purpose of this study is to evaluate the safety and efficacy of A-007, when used to treat high-grade cervical dysplasia.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study. It will randomize patients in a 1:1 ratio to topical cervical treatment with A-007, or placebo gel. Following biopsy confirmation of High Grade Squamous Intraepithelial Lesions (HSIL), women will treat themselves with gel applied to the cervix via an intravaginal applicator. Patients will apply gel once daily for 5 consecutive days of a 28-day cycle for 2 cycles. Women will return to clinic for safety assessments, colposcopy, cytology, and virologic and immunologic testing.

ELIGIBILITY:
Inclusion Criteria:

Patients may be enrolled in the study only if they meet all of the following criteria:

* 18 years of age or older
* The patient or her authorized representative must sign and date an Ethical Review Board-approved informed consent document. All aspects of the protocol must be explained and written informed consent obtained.
* Patients must have histological proof of HSIL (CIN 2/3) disease documented.
* Cervical swabs must test positive for HPV (by Hybrid Capture 2).
* Patients must have a Hb ≥ 9 g/dl, a peripheral WBC ≥ 3000 mm3 and platelet counts ≥ 100,000 mm3.
* Normal hepatic and renal functions - AST and ALT < 2.5 x ULN and creatinine < 1.5 x ULN, respectively.
* Females of childbearing potential must use one of the following birth control methods during the treatment period and 2 weeks thereafter: oral, implantable, injectable contraceptives; abstinence (celibacy). Contraceptive sponges, IUD, spermicides, sponges, condoms, or partner's vasectomy are not acceptable methods of birth control.

Exclusion Criteria:

Patients will be excluded from the study for any of the following preexisting reasons:

* Patients with LSIL (CIN 1) or invasive squamous cell carcinoma (SCC).
* SIL (CIN) involving the endocervix as determined by endocervical curettage, or otherwise not amenable to adequate colposcopic follow-up evaluations, i.e. unsatisfactory colposcopy.
* CIN 3 involving more than two cervical quadrants on colposcopy.
* Patients treated for cervical SIL within the past year.
* Patients with other malignancy (except for non-melanoma skin) within the past 5 years.
* Patients with any active infections (including HIV) other than HPV.
* Patients with known clinically relevant immunological deficiency.
* Concurrent treatment with cytotoxic, radiation, or immuno-stimulative therapy, or with systemic corticosteroids at a dose of > 5 mg/d of prednisone (or its equivalent).
* Participation in another investigational medication trial concurrently or within 30 days, or prior participation in an HPV vaccine trial. Treatment within the last 30 days with a medication that has not received regulatory approval at the time of study entry.
* Concomitant use of topical vaginal medications.
* Significant acute or chronic medical or psychiatric illness that, in the judgment of the Investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study.
* History of allergy or hypersensitivity to cosmetics, toiletries, or other topical or dermatologic products.
* Pregnant or lactating females who are nursing and will not consent to cease nursing.
* Investigators, site personnel directly affiliated with this study, and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Burigo, MD, Principal Investigator — OB/GYN Specialists of the Palm Beaches; Ramon Cestero, MD, Principal Investigator — Arrowhead Regional Medical Center; Paul M Fine, MD, Principal Investigator — Planned Parenthood of Houston & Southeast Texas, Inc.; Keith A Aqua, MD, Principal Investigator — Visions Clinical Research; Steven C Blank, MD, Principal Investigator — Mount Vernon Clinical Research, LLC; Douglas G Young, MD, Principal Investigator — Northern California Research Corp; Allan T Sawyer, MD, Principal Investigator — Hope Research Institute, LLC; Mark H Einstein, MD, Principal Investigator — Montefiore Medical Center-Weiler Division; Robert M Spitz, MD, Principal Investigator — Coastal Connecticut Research, LLC; Thomas A deHoop, MD, Principal Investigator — Greater Cincinnati OB/GYN, Inc.; Lance R Bruck, MD, Principal Investigator — Jacobi Medical Center; Warner K Huh, MD, Principal Investigator — University of Alabama Highlands, Dept. of OB/GYN; Giuseppe Del Priore, MD, Principal Investigator — New York Presbyterian Hospital; Michael A Gold, MD, Principal Investigator — University of Oklahoma Health Sciences Center Dept of OB/GYN; Richard S Guido, MD, Principal Investigator — Magee-Womens Hospital, Dept of OB/GYN & Reproductive Services; Philip E Young, MD, Principal Investigator — IGO Medical Group of San Diego; Daron G. Ferris, MD, Principal Investigator — Augusta University; Cynthia J Goldberg, MD, Principal Investigator — Visions Clinical Research-Tucson; Ana Eduardo, MD, Principal Investigator — Hill Country OB/GYN; Phyllis Gee, MD, Principal Investigator — OB/GYN; Robert Pfeffer, MD, Principal Investigator — Robin Black OGNP, Costa Mesa California; Jonathan A Cosin, MD, Principal Investigator — Medstar Health Research Institute; James A Williams, MD, Principal Investigator — South Carolina Oncology Associates; Vincent A Culotta, Jr, MD, Principal Investigator — East Jefferson OB/GYN; G. Michael Swor, MD, Principal Investigator — Physician Care Clinical Research, LLC.; Garn R Mabey, MD, Principal Investigator — Office of R. Garn Mabey, MD; Martin Martino, MD, Principal Investigator — Lehigh Valley Hospital; Robert Klein, MD, Principal Investigator — Global OB/GYN Centers of Florida; William J Mann, MD, Principal Investigator — Jersey Shore University Medical Center
Locations (29):
- United States (29):
  - University of Alabama Highlands, Dept. of OB/GYN, Birmingham, Alabama
  - Hope Research Institute, LLC, Phoenix, Arizona
  - Visions Clinical Research-Tucson, Tucson, Arizona
  - Northern California Research Corp, Carmichael, California
  - Arrowhead Regional Medical Center, Colton, California
  - Robin Black OGNP, Costa Mesa, California
  - IGO Medical Group of San Diego, San Diego, California
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Visions Clinical Research, Boynton Beach, Florida
  - Global OB/GYN Centers of Florida, Pembroke Pines, Florida
  - Physician Care Clinical Research, LLC., Sarasota, Florida
  - OB/GYN Specialists of the Palm Beaches, West Palm Beach, Florida
  - Mount Vernon Clinical Research, LLC, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - East Jefferson OB/GYN, Metairie, Louisiana
  - Office of R. Garn Mabey, MD, Las Vegas, Nevada
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - New York Downtown Hospital, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center-Weiler Division Dept of OB/GYN & Women's Health, The Bronx, New York
  - Greater Cincinnati OB/GYN, Inc., Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center Dept of OB/GYN, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Magee-Womens Hospital, Dept of OB/GYN & Reproductive Services, Pittsburgh, Pennsylvania
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Hill Country OB/GYN, Austin, Texas
  - Planned Parenthood of Houston & Southeast Texas, Inc., Houston, Texas
  - 4601 Old Shepard Place; Bldg 2, Suite 201, Plano, Texas

REFERENCES:
- [Background] Morgan LR, Thangaraj K, LeBlanc B, Rodgers A, Wolford LT, Hooper CL, Fan D, Jursic BS. Design, synthesis, and anticancer properties of 4,4'-dihydroxybenzophenone-2,4-dinitrophenylhydrazone and analogues. J Med Chem. 2003 Oct 9;46(21):4552-63. doi: 10.1021/jm0301080. PMID 14521417
- [Background] Morgan, LR, Hooper, CL, Rodgers, AH, LoRusso, P, Eilender, DE and Culotta, VA. 4,4'-Dihydroxybenzophenone-2,4-dinitrophenyl-hydrazone (A-007): A CD4+ T-Lymphocyte Modulator Useful in the Treatment of Advanced Cancer. Chemotherapy - accepted 2005.
- [Background] Morgan, LR, Hooper, CL, Rodgers, AH Culotta, V et al. 4,4'-Dihydroxy benzophenone -2,4-dinitrophenylhydrazone (A-007) A Modulator of CD45+ T Lymphocytes in HPV Infected Anogenital Epithelium. In: HPV Vaccines and Immune Therapy, Cambridge, United Kingdom, 2003

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (no treatment)
- A007: Experimental A007
Period: Overall Study
Arm/Group | Placebo | A007
Started | 70 | 77
Treated | 63 | 75
Completed | 61 | 71
Not Completed | 9 | 6
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Pregnancy | 1 | 1
Not completed — non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | A007 | Total
Number analyzed (Participants) | 70 | 77 | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 77 | 147
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28 (6) | 28.7 (7.9) | 28.4 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 77 | 147
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 70 | 77 | 147

OUTCOME MEASURES:

1. Primary Outcome: Pathological Response
Description: Pathological resonse is defined as a patient who regressed from Cervical intraepithelial neoplasia (CIN) 2/3 to normal at the end of 4 months.
Time Frame: baseline and 4 months
Measure: Number; unit: participants
Arm/Group | Placebo | A007
Number analyzed (Participants) | 70 | 77
participants | 20 | 24

2. Secondary Outcome: Local Tolerability and Systemic Safety of A-007 Will be Assessed by Way of CTCAE 3.0.
Time Frame: over the course of the trial
Reporting Status: Not Posted

3. Secondary Outcome: Eradication of Human Papilloma Virus (HPV) Will be Assessed by Way of Cervical Cytology and Swab Collection.
Time Frame: over the course of the trial
Reporting Status: Not Posted

4. Secondary Outcome: Immunologic Parameters B/T Cells Will be Assessed by B/T Cell Profile Collection.
Time Frame: over the course of the trial
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Placebo | A007
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/75
Other Adverse Events (participants affected / at risk) | 2/63 | 5/75
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=63) | A007 (N=75)
Headache (General disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No